CLINICAL TRIAL: NCT01890083
Title: An Exercise Intervention to Prevent Interferon-Induced Depression in Hepatitis C
Brief Title: A Health Intervention to Prevent Depression Hepatitis C Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of eligible patients due to introduction of new drugs for Hepatitis C
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K01MH097847 (NIH)
Record Dates: First submitted 2013-06-05; First posted 2013-07-01 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Hepatitis C; Major Depressive Disorder
Keywords: Hepatitis C; Interferon-alpha; Depression; Major Depressive Disorder; Exercise; Physical Activity
MeSH Terms: conditions — Hepatitis C; Depressive Disorder, Major; Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education (Active Comparator): Participants will three attend heath education sessions per week for 26 weeks.
  Interventions: Behavioral: Health Education
- Exercise (Experimental): Participants will engage in a public health dose of moderate-to-vigorous aerobic exercise for 26 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise
Behavioral: Health Education
  Arms: Health Education

SUMMARY:
Interferon-alpha (IFN-α) is an efficacious treatment for Hepatitis C (HPC); however, IFN-α treatment results in a significant increase in depressive symptoms. The aim of this project is to compare two health interventions (exercise vs. health education) to prevent depression in HPC patients receiving IFN-α. Participants will be recruited from the Clinical Center for Liver Diseases at UT-Southwestern and randomized to 26 weeks of either: aerobic exercise or a health education control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hepatitis C and prescribed IFN-α
* Ability to understand and willingness to provide written informed consent.
* Willing to provide contact information.
* Medical clearance with protocol-defined stress testing (in accordance with American College of Sports Medicine (ACSM) guidelines) from protocol approved medical personnel. Details of guidelines and related testing protocol are provided in the study Manual of Procedures.
* Able to comprehend and communicate in English.

Exclusion Criteria:

* Have a medical condition contraindicating exercise participation
* Are currently physically active - defined as moderate intensity physical activity on 3 or more days per week for the last month
* Have been diagnosed with current Major Depressive Disorder or are currently receiving antidepressant medication treatment (including SSRIs and SNRIs)
* Currently considered a high suicide risk and/or high risk for being unable to complete the study due to the need for psychiatric hospitalization, suicide attempts or suicidality, significant self-mutilation, or other self-injurious or destructive behavior based on the judgment of the site PI, medical personnel, or designee.
* Pregnancy.
* Current psychotic disorder. Other comorbid psychiatric diagnosis that, in the investigator's judgment, will pose a safety issue or make it difficult for the participant to understand or complete the intervention.
* Anticipated circumstances over the 6-month course of the trial that would render the participant unlikely to complete the study in the judgment of the PI or designee.
* Any reason not listed herein yet, determined by the PI, medical personnel, or designee that constitutes good clinical practice and that would in the opinion of the PI, medical personnel, or designee make participation in the study hazardous.
* Are currently enrolled in another research study, and participation in that study contraindicates participation in the current study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Depressive Symptoms over 6 months | Baseline, Weeks 3, 5, 7, 11, 15, 19, 23, 27

SECONDARY OUTCOMES:
Change in Sleep Quality over 6 months | Baseline, Weeks 3, 5, 7, 11, 15, 19, 23, 27
Change in blood biomarkers over 6 months | Baseline, Weeks 3, 5, 7, 11, 15, 19, 23, 27

CONTACTS AND LOCATIONS:
Overall Officials: Chad D Rethorst, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided